CLINICAL TRIAL: NCT07163923
Title: The Role of the MIND Diet in Alzheimer's Disease Patients: A Case-Control Study on Malnutrition and Depression
Brief Title: MIND Diet in Relation to Malnutrition and Depression in AD
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Nurefşan KONYALIGİL ÖZTÜRK, Assist. Prof. Dr., Abant Izzet Baysal University
Other Study IDs: AIBU-BD-NKÖ-01
Record Dates: First submitted 2025-08-28; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease (AD); Healthy Controls Group - Age and Sex-matched
Keywords: Alzheimer disease; Depression; Diet; Malnutrition
MeSH Terms: conditions — Alzheimer Disease; Depression; Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer's Disease Patients: Participants diagnosed with Alzheimer's disease according to established clinical criteria. Evaluated for malnutrition and depression status. No intervention was applied.
- Healthy Controls: Age- and sex-matched individuals without Alzheimer's disease. Evaluated for malnutrition and depression status. No intervention was applied.

SUMMARY:
The aim of this study was to examine the association between depression, malnutrition, and the Mediterranean-Dietary Approaches to Stop Hypertension Diet Intervention for Neurodegenerative Delay (MIND) diet in Alzheimer's disease patients. This study included 30 patients with Alzheimer's disease (AD) and 30 healthy controls. A questionnaire form including sociodemographic characteristics was applied to the individuals. In addition, anthropometric measurements, biochemical parameters, nutritional status (Food Frequency Questionnaire (FFQ), Mini Nutritional Assessment-Short Form (MNA-SF), Geriatric Nutritional Risk Index (GNRI) and MIND diet scores) and mental health status (Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI)).

DETAILED DESCRIPTION:
Significant progress has been made in understanding the neurobiological basis and treatment approaches for Alzheimer's disease (AD) and depression; however, the biological link between these two disorders has not yet been fully elucidated. A deeper understanding of this relationship could contribute to the development of more effective strategies for the prevention and treatment of both conditions. In this context, lifestyle-based interventions, such as nutrition, which have been shown to support cognitive health, emerge as a potential preventive and therapeutic approach. Therefore, the aim of this study was to examine the relationship between depression, malnutrition, and the Mediterranean-Dietary Approaches to Stop Hypertension Diet Intervention for Neurodegenerative Delay (MIND) diet in individuals with AD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 60 years.
* Diagnosed with Alzheimer's disease (AD) (for AD group)
* Able to communicate with themselves or their companions
* Healthy volunteers without systemic or neurological diseases (for control group)
* Matching criteria: Age, gender, smoking status, and alcohol use

Exclusion Criteria:

* Chronic inflammatory diseases
* Schizophrenia
* Bipolar disorder
* Amputations
* Neoplastic disorders
* End-stage liver disease
* End-stage kidney disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was planned as a case-control study. The study was conducted on healthy individuals with AD who were admitted to Bolu Abant İzzet Baysal University Training and Research Hospital Neurology Outpatient Clinic and volunteered to participate in the study. In the study, according to the 5% significance level (α = 0.05), 80% statistical power (1-β = 0.80) and sample size calculation for two groups (AD and control group), it was determined that at least 30 individuals should be included in each group in order to detect a medium-large effect size (Cohen's d ≈ 0.66). Therefore, 30 AD and 30 healthy individuals (control group) who volunteered to participate in the study were included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire Form | 4 months
  Sociodemographic characteristics of the individuals (age, gender, smoking and alcohol use, constipation status, swallowing-chewing problem) were questioned.
Body weight (BW) | 4 months
  BW was measured using a calibrated digital scale placed on a flat, tiled surface. The scale was sensitive to 100 grams.
Height | 4 months
  Height was measured using a stadiometer with the participant's head positioned in the Frankfort plane and feet placed together.
Waist Circumference (WC) | 4 months
  WC was measured at the midpoint between the lowest rib and the iliac crest (cristal point) using a flexible measuring tape.
Hip Circumference (HC) | 4 months
  HC was measured at the widest point of the hips using a flexible measuring tape.
Body Mass Index (BMI) | 4 months
  BMI was calculated by dividing body weight (in kilograms) by the square of height (in meters): BMI = weight (kg) / height² (m²).
Fasting Blood Glucose | 4 months
  Fasting blood glucose was measured using standard laboratory techniques during routine outpatient visits.
Triglycerides | 4 months
  Triglyceride levels were measured via fasting blood samples analyzed in the outpatient clinic laboratory.
LDL-Cholesterol | 4 months
  LDL-cholesterol was measured from fasting serum samples using standard enzymatic colorimetric methods.
Total Cholesterol | 4 months
  Total cholesterol was measured using routine biochemical analysis in a certified laboratory.
Albumin | 4 months
  Serum albumin levels were measured using routine laboratory procedures in outpatient visits.
Vitamin D | 4 months
  Serum vitamin D (25(OH)D) levels were assessed using chemiluminescence immunoassay methods in the outpatient clinic laboratory.
Folic Acid | 4 months
  Serum folic acid levels were measured using standard automated immunoassay techniques.immunoassay methods in the outpatient clinic laboratory.
Vitamin B12 | 4 months
  Serum vitamin B12 concentrations were measured using automated chemiluminescent immunoassay.immunoassay methods in the outpatient clinic laboratory.
Food Frequency Questionnaire | 4 months
  The foods consumed by individuals in the last month were evaluated across seven different groups, including five basic food groups (meat and meat products, milk and dairy products, bread and grains, vegetables and fruits, sugar and fats), beverages, and fast food. Participants were asked how often they consumed foods and beverages in these groups; responses were collected using the following options: "every meal," "every day," "5-6 days a week," "3-4 days a week," "1-2 days a week," "once every 15 days," "once a month," and "never." To determine the average daily consumption amounts based on consumption frequency, the following coefficients were used: 3 for "every meal," 1 for "every day," 0.7855 for "5-6 times a week," 0.498 for "3-4 times a week," 0.2145 for "1-2 times a week," 0.067 for "every 15 days," and 0.033 for "once a month."
MIND diet compliance score | 4 months
  It includes a total of 15 different food groups, ten groups that protect brain health and five groups that harm brain health. By examining the Food Frequency Questionnaire of individuals, the amount of consumption of foods belonging to these 15 groups was divided into portions and evaluated in accordance with the scoring. It is scored between 0-15 and there is no cut-off point for determining compliance with the Mediterranean-Dietary Approaches to Stop Hypertension Diet Intervention for Neurodegenerative Delay (MIND) diet. It has been reported that the higher the score, the higher the compliance with the MIND diet. The Food Frequency Questionnaire of the items reflecting each MIND diet component were quantified in terms of how many days per week individuals consumed the food item.
Geriatric Nutritional Risk Index (GNRI) | 4 months
  It was first introduced to evaluate the nutritional status of elderly, bedridden care patients. GNRI is calculated using height, weight and serum albumin values of the patients. GNRI [1.489 x albumin (g/l)] + [ 41.7 x (body weight / ideal body weight)]. According to the GNRI results, they are divided into four groups. Malnutrition grades are grouped as GNRI<82; severe malnutrition, moderate malnutrition between 82-92, mild malnutrition between 92-98, and no risk for malnutrition above 98.
Mini Nutritional Assessment-Short Form (MNA-SF) | 4 months
  It is a screening tool used to evaluate malnutrition in elderly individuals. The tool includes six items that assess various factors such as appetite changes, unintentional weight loss over the past three months, neuropsychological issues, presence of psychological stress or acute illness, mobility, and BMI. Based on the total score, individuals are categorized into three nutritional status groups: 0-7 points: Malnourished (indicating nutritional deficiency), 8-11 points: At risk of malnutrition, 12-14 points: Normal nutritional status.
Beck Depression Inventory (BDI) | 4 months
  The BDI was developed to measure behavioral symptoms of depression in adolescents and adults. The inventory was revised to remove repetitive statements describing severity levels and to ask individuals to assess not only their mood on that day but also their mood over the past week. The scores obtained from the inventory are classified as follows to determine the severity of depression: 0-9 points: Minimal depression, 10-16 points: Mild depression, 17-29 points: Moderate depression, 30-63 points: Severe depression.
Beck Anxiety Inventory (BAI) | 4 months
  It was originally developed to assess the intensity and frequency of anxiety symptoms reported by individuals. This self-assessment tool comprises 21 items, each rated on a scale from 0 (not at all) to 3 (severely). The total possible score ranges between 0 and 63, and the anxiety level is interpreted based on the total score as follows: 0-7: Minimal anxiety, 8-15: Mild anxiety, 16-22: Moderate anxiety, 23-63: Severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nurefşan Konyalıgil Öztürk, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Health Sciences, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No